CLINICAL TRIAL: NCT00801008
Title: Exercise and Relaxation Intervention for Young Adult Cancer Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Miriam Hospital (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other)
Responsible Party: Principal Investigator, Carolyn Rabin, Assistant Professor (Research), The Miriam Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-091-01-CPPB; MRSG-09-091-01-CPPB
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Cancer
Keywords: young adult; cancer; exercise; relaxation
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise and Relaxation Intervention (Experimental): Participants in this arm will receive a 12 week exercise and relaxation intervention
  Interventions: Behavioral: Exercise and relaxation intervention
- Wait List Control Condition (No Intervention): Participants in this arm will be offered the exercise and relaxation intervention after a 12 week delay.
  Interventions: Behavioral: Exercise and relaxation intervention

INTERVENTIONS:
Behavioral: Exercise and relaxation intervention — Comparison of an exercise and relaxation intervention to a wait-list control condition

SUMMARY:
The purpose of this study is to develop an exercise and relaxation program for young adults (age 18 to 39) who have completed their treatment for cancer.

DETAILED DESCRIPTION:
There is evidence that cancer diagnosis and treatment during young adulthood puts survivors at risk for a number of medical and psychosocial difficulties including cardiovascular disease, second cancers and psychological distress. The proposed research is aimed at developing a physical activity and relaxation intervention for young adult cancer survivors in order to address some of their medical and psychosocial risks. The objective of the study is to pilot test a 12-week physical activity and relaxation intervention in this population. We hypothesize that the intervention will be feasible for and acceptable to young adult cancer survivors. We also hypothesize that the intervention group will demonstrate increased levels of physical activity, improved mood and reduced fatigue relative to the wait list control group at the 12-week and 24-week follow-up assessments; statistically significant differences may not be found due to the small sample size, however. In addition, we will conduct exploratory tests of intervention effects on fitness, flexibility, body mass, and waist circumference. Sixty participants will be recruited for the pilot study. Participants will be randomly assigned to receive a 12-week physical activity and relaxation intervention or to a wait list control group. Intervention group participants will receive 12 weeks of behavior change counseling, based on the Transtheoretical Model and Social Cognitive Theory, to help them adopt a program of brisk walking and learn mindfulness meditation. They will also be given access to an online discussion group. Participants in both arms of the study will be assessed at baseline, 12 weeks, and 24 weeks. Following the 24-week assessment, wait list control participants will offered the 12-week intervention and one additional assessment (i.e., at 36 weeks). Data will be collected on intervention feasibility (e.g., number of counseling sessions delivered) and acceptability (e.g., general satisfaction ratings). ANCOVAs will be used to conduct preliminary tests of intervention effects (e.g., on physical activity, mood, and fatigue).

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 39
* diagnosed with any form of cancer (except non-melanoma skin cancer)
* diagnosed between age 18 and 39 in the past 10 years
* completed all surgery, chemotherapy and radiation therapy
* currently in a cancer remission
* able to speak and write English fluently
* sedentary (i.e., not regularly physically active)
* not currently engaging in a relaxation strategy
* score above a cutoff on a fatigue screener

Exclusion Criteria:

* the intention to get pregnant
* the presence of a known medical condition or history of severe psychiatric illness that would make participation dangerous or very difficult

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-07; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility measure: number of counseling sessions delivered | 12 weeks
Acceptability measure: response to the item "In general how satisfied were you with the intervention?" | 12 weeks

SECONDARY OUTCOMES:
Minutes of moderate-intensity activity on Seven Day PAR | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Rabin, PhD, Principal Investigator — The Miriam Hospital
Locations (1):
- Miriam Hospital, Providence, Rhode Island, United States